CLINICAL TRIAL: NCT03515577
Title: Prospective Single Center Trial to Compare 68Ga-PSMA-11 and Axumin PET/CT (18F-Fluciclovine) for Restaging Prostate Cancer Patients With Biochemical Recurrence After Radical Prostatectomy
Brief Title: Gallium Ga 68-labeled PSMA-11 PET/CT and Fluciclovine F18 PET/CT in Imaging Participants With Recurrent Prostate Cancer After Surgery
Acronym: PSMA vs AXUMIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-001885; NCI-2018-00546 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-001885 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2018-04-20; First posted 2018-05-03 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2019-06

CONDITIONS: Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluciclovine F-18; gallium 68 PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Diagnostic ([68]Ga-PSMA-11 PET/CT, Axumin PET/CT) (Experimental): Participants receive (68)Ga-PSMA-11 IV and 60-90 minutes later, undergo PET/CT imaging over 3 hours. Participants also undergo best standard of care Axumin PET/CT within 2 weeks before or after (68)Ga-PSMA-11 PET/CT.
  Interventions: Procedure: Computed Tomography; Drug: Fluciclovine F18; Drug: Gallium Ga 68-labeled PSMA-11; Other: Laboratory Biomarker Analysis; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Drug: Fluciclovine F18 — Given fluciclovine F18
  Other Names: (18F)Fluciclovine; (18F)GE-148; 18F-Fluciclovine; [18F]FACBC; Anti-(18f)FABC; Anti-1-Amino-3-[18F]Fluorocyclobutane-1-Carboxylic Acid; Anti-[18F] FACBC; Axumin; Fluciclovine (18F); FLUCICLOVINE F-18; GE-148 (18F); GE-148 F-18
Drug: Gallium Ga 68-labeled PSMA-11 — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA-11; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga-68 labeled PSMA-11; Gallium Ga 68 PSMA-11; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; PSMA-HBED-CC GA-68
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase II trial compares how well gallium 68-labeled PSMA-11 positron emission tomography/computed tomography (PET/CT) works compared to fluciclovine F18 PET/CT in imaging participants with prostate cancer after surgery that has come back. PET is an established imaging technique that uses small amounts of radioactivity and CT images provide an exact outline of organs and potential inflammatory tissue where it occurs in the body. Diagnostic procedures, such as PET/CT with gallium 68-labeled PSMA-11, may work better than PET/CT with fluciclovine F18 in helping find out how far the prostate cancer has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the detection rates of gallium 68-labeled PSMA-11 ([68]Ga-PSMA-11) PET/CT and fluciclovine F18 (Axumin) PET/CT for the identification of tumor location(s), by patient and region based analysis.

SECONDARY OBJECTIVES:

I. Detection rate on a per-patient basis of (68)Ga-PSMA-11 PET/CT and Axumin PET/CT, stratified by prostate-specific antigen (PSA) value (0.2 - < 0.5; 0.5 - < 1.0; 1.0 - < 2.0).

II. Sensitivity and positive predictive value (PPV) on a per-patient basis, of (68)Ga-PSMA-11 PET/CT and Axumin PET/CT for the detection of tumor location(s), confirmed by histopathology/biopsy and/or clinical and conventional imaging follow-up.

III. Agreement among the readers, separate for (68)Ga-PSMA-11 PET/CT versus Axumin PET/CT.

OUTLINE:

Participants receive (68)Ga-PSMA-11 intravenously (IV) and 60-90 minutes later, undergo PET/CT imaging over 3 hours. Participants also undergo best standard of care Axumin PET/CT within 2 weeks before or after (68)Ga-PSMA-11 PET/CT.

After completion of the PET/CT scan, participants are followed up between 1 and 3 days and up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven prostate cancer (PCa)
* Radical prostatectomy as definitive treatment for PCa
* Proven biochemical recurrence as defined by American Urological Association (AUA) recommendation: PSA greater than or equal to 0.2 ng/mL measured more than 6 weeks after radical prostatectomy
* PSA values ranging from 0.2 ng/mL to 2 ng/mL
* No prior salvage therapies (including salvage radiotherapy and/or salvage lymph node dissection)
* Axumin PET/CT scan already performed or scheduled as best standard of care procedure for suspected disease relapse within 2 weeks before or after intended 68Ga-PSMA-11 PET/CT
* Karnofsky performance status of ≥ 50 (or Eastern Cooperative Oncology Group (ECOG)/World Health Organization [WHO] equivalent)
* Ability to understand a written informed consent document and the willingness to sign it

Exclusion Criteria:

* Any change in prostate cancer treatment between Axumin and 68Ga-PSMA PET/CT scan
* Unable to lie flat, still or tolerate a PET scan

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Gallium 68-labeled PSMA-11 ([68]Ga-PSMA-11) and fluciclovine F18 (Axumin) detection rates | Up to 15 months: through data analysis completion (anonymized central imaging read), an estimation of 3 months after enrollment completion.
  Will compare rates for the identification of tumor location(s), assessed by patient and region based analysis. This will be calculated and reported along with the corresponding two-sided 95% confidence intervals. The confidence intervals will be constructed using the Wilson score method. Detection rate in the per-participant analysis is defined as number of participants with PET positive disease, independent of pathology or imaging/clinical follow-up. Detection rate in the per-region analysis is defined as number of regions (prostate bed, pelvic lymph-nodes, extra-pelvic lymph-nodes, bone metastases, other soft tissue) resulted PET positive, independent of pathology or imaging/clinical follow-up.

SECONDARY OUTCOMES:
Detection rates on a per-patient basis of 68^Ga-PSMA-11 PET and Axumin PET | Up to 1 year after completion of PET/CT with 68^Ga-PSMA-11
  This will be stratified by prostate-specific antigen (PSA) value (0.2 - < 0.5, 0.5 - < 1.0, 1.0 - < 2.0, 2.0 - < 5.0, ≥ 5.0) and will be summarized in tabular format and compared between PSA using chi-square analysis. Detection rate is defined as number of participants with PET positive disease, independent of pathology, imaging or clinical follow-up.
Sensitivity and PPV by-participant and region-based analysis of 68^Ga-PSMA-11 PET and Axumin PET for detection of tumor location(s) | Up to 1 year after completion of PET/CT with 68^Ga-PSMA-11
  The sensitivity and positive predictive values (PPV) will be calculated and reported along with the corresponding two-sided 95% confidence intervals. The confidence intervals will be constructed using the Wilson score method. Only participants having histopathology/biopsy and/or clinical and conventional imaging follow-up will be analyzed
Inter-observer (reader) agreement | Up to 15 months: through data analysis completion (anonymized central imaging read), an estimation of 3 months after enrollment completion.
  Agreement will be calculated separately for 68^Ga-PSMA-11 PET/CT versus Axumin PET/CT. For binary data, agreement among central readers will be evaluated using Fleiss' k. For non-binary data with more than ten observations, agreement among central readers will be evaluated by interclass correlation coefficient (ICC). Ninety-five percent confidence intervals (CIs) will be reported for k and ICC values. Interpretation of k and ICC will be based on a classification provided by Landis and Koch: 0.0, poor; 0.0-0.20, slight; 0.21-0.40, fair; 0.41-0.60, moderate; 0.61-0.80, substantial; 0.81-1.00, almost-perfect reproducibility.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Czernin, M.D., Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Result] Calais J, Ceci F, Eiber M, Hope TA, Hofman MS, Rischpler C, Bach-Gansmo T, Nanni C, Savir-Baruch B, Elashoff D, Grogan T, Dahlbom M, Slavik R, Gartmann J, Nguyen K, Lok V, Jadvar H, Kishan AU, Rettig MB, Reiter RE, Fendler WP, Czernin J. 18F-fluciclovine PET-CT and 68Ga-PSMA-11 PET-CT in patients with early biochemical recurrence after prostatectomy: a prospective, single-centre, single-arm, comparative imaging trial. Lancet Oncol. 2019 Sep;20(9):1286-1294. doi: 10.1016/S1470-2045(19)30415-2. Epub 2019 Jul 30. PMID 31375469